CLINICAL TRIAL: NCT04470765
Title: Transcutaneous Tibial Nerve Stimulation: the ZIDA Device
Brief Title: Transcutaneous Tibial Nerve Stimulation: the ZIDA Device Equivalence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Exodus Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-9050 v1.0.6
Record Dates: First submitted 2020-07-07; First posted 2020-07-14 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Overactive Bladder; Urge Incontinence; Urinary Incontinence; Urinary Frequency More Than Once at Night
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence; Nocturia

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized, single-blind, placebo-controlled study of 50 subjects divided into two groups, with one group having the active ZIDA device treatment once weekly at home, and one group having a sham ZIDA device (non-treatment) once weekly at home, for a duration of 12 weeks for both groups. Subjects will be called by a research member weekly to report their weekly treatment and any complications during the 12-week treatment period. A phone call assessment will be conducted during week-6 period. Subjects will complete a final phone-call assessment at the end of the week-12 period.
  This clinical investigation is being conducted in accordance with 21 CFR Parts 50, 54, 56, and abbreviated 21 CFR 812 regulations, International Conference on Harmonization Good Clinical Practice (ICH GCPs), applicable local regulations and Institutional Review Board (IRB) requirements.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A third party will be assigned to label the devices prior to distribution to the study center. The 3rd party will maintain blinding of the device labelling/ assignment codes until the trial completion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Treatment (Active Comparator): Active Zida device to be delivered for use by patient
  Interventions: Device: Zida
- Sham Treatment (Sham Comparator): Identical Sham device to be delivered for use by patient
  Interventions: Device: Zida

INTERVENTIONS:
Device: Zida — Transcutaneous Tibial Nerve Stimulation

SUMMARY:
Tibial nerve stimulation (TNS) has been shown to be an effective alternative for the management of the overactive bladder (OAB). Transcutaneous Tibial Nerve Stimulation (TTNS) uses a series of regular electrical pulses to stimulate the tibial nerve. Numerous studies have positively shown the efficacy of this treatment. These studies have included multicentric, double-blind, randomized sham-controlled study of patients with idiopathic OAB. , . In 2013 the British National Institute for Health and Care Excellence (NICE) guidance has added TTNS as a second-line option for the management of female urinary incontinence , .

In reality, the vast majority of patients treated using tibial nerve receive treatment percutaneously (PTNS) by inserting a needle into their lower leg. PTNS requires 12 visits to a physician's office and a painful treatment experience. From a physician's perspective PTNS is resource intensive in terms of time, financial and staff commitments. As a result, PTNS is often not a feasible option from the point of view of health care delivery. Moreover, the treatment may not be an option for patients whose schedule or ability to travel is limited. These issues are exacerbated for those with disabilities requiring special transport arrangements and who have trouble committing to 12 expensive and long trips to receive treatment. Additionally, 8% of patients who undergo PTNS complain of adverse effects which include pain, bruising, tingling or bleeding at the insertion site of the 34-gauge needle. As a direct result of these limitations long-term follow up studies of patients undergoing PTNS treatment show poor compliance to PTNS over time .

Non-invasive, homecare TTNS devices such as the ZIDA Wearable Neuromodulation System are on the cusp of achieving regulatory clearance. TTNS, stimulates transcutaneously at a home-based setting and at least one study has explored the efficacy of this treatment method . Early results have demonstrated improvements in OAB symptom scores and urodynamic parameters . So far, these studies have employed standard commercial TENS devices (transcutaneous electrical nerve stimulation). These studies have used a variety of treatment frequencies to stimulate the tibial nerve at frequencies between 10 to 40 Hz, patient have been advised which pre-determined stimulation settings can be used for home care treatment. Commercial TENS devices limit mobility of patients during the time that the nerve is being stimulated.

DETAILED DESCRIPTION:
The ZIDA device uses a series of regular electrical pulses to stimulate the tibial nerve for the management of overactive bladder by a patient in the home setting. The most common potential risk and complication associated with the ZIDA device are discomfort and pain (including throbbing pain) at, or near the stimulation site, including the patient's lower leg and foot; Redness/inflammation at, or near, the stimulation site; Numbness of toes. This study is designed to exclude those subjects who may be at risk for known and unknown complications. No other complications have been reported and there are no new or other expected complications or risks expected in this clinical study, making the safety profile of the ZIDA no greater than that of other tibial nerve stimulator products that are commercially used for treatment of overactive bladder.

As mentioned above, the ZIDA device has a low potential for risks and complications. Therefore, the study Sponsor and Principle Investigator have determined that through their participation in this clinical study, the study subjects will be exposed to no new risks compared to the risks of devices currently available for similar intended uses. Specifically, the proposed study of ZIDA meets the definition of an NSR (nonsignificant risk) study for the following reasons:

* ZIDA is NOT intended as an implant
* ZIDA is NOT purported or represented to be for use supporting or sustaining human life
* ZIDA does NOT present a potential for serious risk to the health, safety or welfare of a subject
* ZIDA has a very low safety risk profile.
* The study will be conducted by investigational centre and investigators with experience and expertise and sufficient staff to provide quality care to subjects requiring treatment of an overactive bladder.
* The study was designed to mitigate any potential unknown risk through the eligibility criteria, subject selection and training on the ZIDA device.

As addressed above, the ZIDA device does NOT otherwise present a potential for serious risk to the health, safety or welfare of a subject and meets the definition of a NSR study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give informed consent for participation in the trial.
* Subject is Male or Female, aged 21 years or older.
* Subject has been diagnosed with overactive bladder (OAB).

  o Subject eligibility is based on meeting the criteria for an OAB, defined by the International Continence Society as an average urinary frequency: ≥8 voids and ≥1 urgency episode (with or without incontinence) per 24 hours .
* Subject has clinically acceptable laboratory results within 30 days of enrolment Urinalysis: Dipstick

Acceptable results:

* pH - results not relevant
* Specific gravity - results not relevant
* Glucose - results not relevant
* Ketones - results not relevant
* Nitrites - normal
* Leukocyte esterase (leukocytes) - normal
* Bilirubin - results not relevant
* Urobilirubin - results not relevant
* Blood - normal
* Protein - results not relevant If the urinanalysis is normal no further laboratory studies are indicated. If the urinanalysis abnormal then patient should not be admitted into trial.
* Subject has a score of 60 or higher on the Incontinence impact questionnaire-OAB-q Short Form, 4-week recall.
* In the Investigator's opinion, Subject is able and willing to comply with all trial requirements, including the use of the investigational device in a home setting.
* Subject is willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* The Subject may not enter the trial if ANY of the following apply:

  * Female Subject who is pregnant, lactating or planning pregnancy during the course of the trial.
  * Administration of intravesical injection of botulinum toxin within 36 months of study enrolment.
  * A treatment within the previous year of neuromodulation (TNS or sacral neuromodulation) for OAB.
  * Subject with sensory loss in the gaiter region (cutaneous sensation to nociception was assessed in the lower limb).
  * Presence of urinary tract infection or any other documented lower urinary tract (LUT) pathology.
  * Subject with pacemakers or implantable defibrillators
  * Subject who have participated in another research trial involving an investigational product in the past 12 weeks.
  * Subjects with neurological disease
  * Subject on antimuscarinic medications for OAB who have not gone through a 2-week run-in washout period during which time medications were discontinued.
  * Subject is a prisoner or is mentally incompetent.
  * Subject has inflamed, infected or otherwise compromised skin in the area of treatment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical success rate of Zida device in treating OAB | 12 weeks
  The primary efficacy endpoint will be analysed for the FAS population. The primary endpoint is the difference in treatment success between the Zida arm and the sham arm. Treatment success is defined as at least a 30% reduction in the frequency of daytime, night time, or moderate/severe/incontinence voids from baseline to week 12 from an average of the three day ICIQ bladder diary. A chi square test will be used to compare the clinical success rates between the treatment arms.

SECONDARY OUTCOMES:
Impact of Zida device on patient quality of life as measured by quality of life questionnaire. | 12 weeks
  This secondary endpoint is the difference in change in QOL score from baseline to week 12 between the Zida arm and the sham arm.
Frequency of daily voids | 12 weeks
  This secondary efficacy endpoint is a comparison the change from baseline to week 12 in frequency of daily (daytime and nighttime) voids in the ZIDA arm from an average of the three day ICIQ bladder diary to the reported frequency.
Frequency of moderate/severe/incontinence voids | 12 weeks
  This secondary efficacy endpoint is a comparison the change from baseline to week 12 in frequency of moderate/severe/incontinence voids in the ZIDA arm from an average of the three day ICIQ bladder diary to the reported frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- Miami Medical Consultants, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cava R, Orlin Y. Home-based transcutaneous tibial nerve stimulation for overactive bladder syndrome: a randomized, controlled study. Int Urol Nephrol. 2022 Aug;54(8):1825-1835. doi: 10.1007/s11255-022-03235-z. Epub 2022 May 27. PMID 35622269